CLINICAL TRIAL: NCT05456464
Title: Fatigue and Sleep Quality in Multiple Sclerosis Patients: Does Reiki Application Affect?
Brief Title: Fatigue and Sleep Quality in Multiple Sclerosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Sabahattin Zaim University (Other)
Responsible Party: Principal Investigator, Zülfünaz ÖZER, Investigator, Istanbul Sabahattin Zaim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 6812
Record Dates: First submitted 2022-07-05; First posted 2022-07-13 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Multiple Sclerosis
Keywords: Reiki; Fatigue; Sleep quality; Nursing
MeSH Terms: conditions — Multiple Sclerosis; Fatigue; Sleep Initiation and Maintenance Disorders | interventions — Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: The research will be conducted as a randomized, experimental study with a pretest-posttest control group.
Who Masked: Participant
Masking Description: Reiki and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reiki (Experimental): The researcher, a second-degree Reiki therapist, performed the Reiki therapy. Patients were told to lie comfortably on their backs after they were informed about the therapy. Each of the 7 Reiki hand positions was applied sequentially. Each of the hand positions took 2-3 minutes, requiring 30-40 minutes in total.
  Interventions: Other: Reiki
- Control group (No Intervention): Routine maintenance will be applied

INTERVENTIONS:
Other: Reiki — Reiki is applied touching the energy centers of the body (chakras). There are seven main and many small chakras on a body. Chakras are located on the front and back sides of the body in a vertical line that runs along the middle of the body in humans. A complete Reiki therapy includes all the chakras and organs.
  Arms: Reiki

SUMMARY:
This study was planned to examine the effect of reiki application on fatigue and sleep quality in patients with multiple sclerosis.

DETAILED DESCRIPTION:
Fatigue and Sleep Quality in Multiple Sclerosis Patients: Does Reiki Application Affect?

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Volunteering to participate in the research
* Having the ability to use technological tools
* Not using Reiki and similar integrative treatment methods
* Not having a verbal communication disability (hearing and speaking)
* Not having a diagnosed psychiatric disorder
* Patients who have been treated for MS for more than three months
* Having a scale score of >5 on the Piper Fatigue Scale
* A score of >5 on the Pittsburgh Sleep Quality Scale

Exclusion Criteria:

* None

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
The Piper Fatigue Scale | At the end of Session 1(In the first week, the first session will be face-to-face and the other sessions will be online for 4 days. 1 online session will be given on the first day of the 2nd, 3rd and 4th week. A total of 7 sessions of Reiki will begiven)
  It is a 22-item scale that measures four subscales: behavior (6 items), affect (5 items), sensory (5 items), and cognition/mood (6 items). Each item has 11 response categories on a 0-10 metric with verbal descriptors anchoring the endpoints. Each subscale is scored individually and then aggregated together for an overall score, with higher scores reflecting more fatigue.
The Piper Fatigue Scale | At the end of Session 7(In the first week, the first session will be face-to-face and the other sessions will be online for 4 days. 1 online session will be given on the first day of the 2nd, 3rd and 4th week. A total of 7 sessions of Reiki will begiven)
  It is a 22-item scale that measures four subscales: behavior (6 items), affect (5 items), sensory (5 items), and cognition/mood (6 items). Each item has 11 response categories on a 0-10 metric with verbal descriptors anchoring the endpoints. Each subscale is scored individually and then aggregated together for an overall score, with higher scores reflecting more fatigue.
Pittsburgh Sleep Quality Index (PSQI) | At the end of Session 1(In the first week, the first session will be face-to-face and the other sessions will be online for 4 days. 1 online session will be given on the first day of the 2nd, 3rd and 4th week. A total of 7 sessions of Reiki will begiven)
  The PSQI is a valid and consistent survey comprising of 19 questions to assess quality and amount of sleep and the existence of a sleep disorder and its level in the previous month. The scale was adapted into the Turkish language by Agargün et al. (1996). The scale consists of seven components that assess patients subjective sleep quality, sleep delay, use of sleeping medication and disfunction in daily activities. Each item scores in the range 0-3 points and the total score of the seven components gives the total PSQI score. The total score has a value between 0-21 and a high total score demonstrates a poor quality of sleep. A total PSQI score which is ≤5 indicates "good sleep", and a score which is >5 indicates "poor sleep"
Pittsburgh Sleep Quality Index (PSQI) | At the end of Session 7(In the first week, the first session will be face-to-face and the other sessions will be online for 4 days. 1 online session will be given on the first day of the 2nd, 3rd and 4th week. A total of 7 sessions of Reiki will begiven)
  The PSQI is a valid and consistent survey comprising of 19 questions to assess quality and amount of sleep and the existence of a sleep disorder and its level in the previous month. The scale was adapted into the Turkish language by Agargün et al. (1996). The scale consists of seven components that assess patients subjective sleep quality, sleep delay, use of sleeping medication and disfunction in daily activities. Each item scores in the range 0-3 points and the total score of the seven components gives the total PSQI score. The total score has a value between 0-21 and a high total score demonstrates a poor quality of sleep. A total PSQI score which is ≤5 indicates "good sleep", and a score which is >5 indicates "poor sleep"

CONTACTS AND LOCATIONS:
Overall Officials: Zülfünaz Özer, PhD, Study Director — Istanbul Sabahattin Zaim University
Locations (1):
- Istanbul Sabahattin Zaim University, Faculty of Health Sciences, Istanbul, Güneydoğu Anadolu Bölgesi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Demir M, Can G, Kelam A, Aydiner A. Effects of Distant Reiki On Pain, Anxiety and Fatigue in Oncology Patients in Turkey: A Pilot Study. Asian Pac J Cancer Prev. 2015;16(12):4859-62. doi: 10.7314/apjcp.2015.16.12.4859. PMID 26163604